CLINICAL TRIAL: NCT02003326
Title: Strain and Blood Inflammatory Markers as Prognostic Tools for ARDS AMIS (ARDS - Markers of Inflammation - Strain)
Acronym: AMIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low number of patients enrolled
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13AOI07
Record Dates: First submitted 2013-11-07; First posted 2013-12-06 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inflammatory markers (Other): All patients with inclusion criteria (ARDS moderate and severe: Berlin definition) and absence of non inclusion criteria will have a broncho alveolar wash at day 0 and blood sample every three day to measure inflammatory markers. All patients will receive protective ventilation with low tidal volume and pressures limited (Pplat <30cmH2O). End-Expiratory Lung Volume and strain will be measured every 6 hours from the inclusion to the extubation.
  Interventions: Other: Inflammatory markers

INTERVENTIONS:
Other: Inflammatory markers

SUMMARY:
The objective is determine the strain measured at the bedside could be a dynamic prognostic marker of during Acute respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
Nowadays ARDS severity, and therapeutic efficiency are evaluated using PaO2/FiO2 ratio. Inflammation is a cornerstone of ARDS and the ratio is not a sufficiently accurate tool to predict the evolution of ARDS. A reproducible marker would be helpful to adapt the therapeutics and maybe limit their deleterious effects.

The investigators made the hypothesis that patients moderate to severe ARDS (comparable PaO2/FiO2 ratio) with a higher strain may have higher inflammation.

Moderate/severe ARDS will be ventilate with protective ventilation (low tidal volume and PEEP set to limit plateau pressure under 30cmH2O). Markers of inflammation will be measured in the broncho Alveolar Lavage the first day and in the blood the following days. Strain will be measured at the bedside using the nitrogen washout-washin. Markers of inflammation and strain will be analysed with ventilatory and oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe ARDS (Berlin Definition)
* Acute beginning <1 week
* PaO2/FiO2 ratio ≤ 200 after 24h mechanical ventilation with PEEP≥5cmH2O
* Bilateral opacities on chest X-ray
* Respiratory failure not fully explain by cardiac failure or fluid overload
* Informed consent signed by the next of kin and secondarily by the patient when awake
* Patient with social insurance

No Inclusion criteria

* Age < 18
* Pregnancy a pregnancy test will be done to women of childbearing age
* Chronic obstructive pulmonary disease
* Severe hypoxemia PaO2/FiO2 <50% with high PEEP
* Immunosuppressive treatment
* Immunodeficiency onco-hematology, HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
measure of the number of hours spent with a PaO2/FiO2 ratio under 200mmHg | until the 13th day
  measure of the number of hours spent with a PaO2/FiO2 ratio under 200mmHg : day 0,1,2,4,6,13

SECONDARY OUTCOMES:
Mortality at D28 | at the 28th day
  Verify if the patient is death at the 28th day
Ventilatory free days at D28 | at the 28th day
  To determine if the patient is free ventilatory at the 28th day

CONTACTS AND LOCATIONS:
Overall Officials: Jean DELLAMONICA, MD, Principal Investigator — CHU de Nice Hôpital de l'Archet
Locations (1):
- Réanimation Médicale CHU de Nice - Hôpital de l'Archet, Nice, France